CLINICAL TRIAL: NCT00169013
Title: Gabapentin in the Prevention of Phantom Limb Pain
Brief Title: Gabapentin in Phantom and Stump Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Danish Pain Research Center (Other)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Gabapentin2002
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2024-08-09 (Actual); Status verified 2007-04

CONDITIONS: Amputation of Lower Limb
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Gabapentin

SUMMARY:
To investigate whether gabapentin can prevent phantom and stump pain after amputation.

ELIGIBILITY:
Inclusion Criteria:

1. Amputation of crus or femur

Exclusion Criteria:

1. Patients who cannot cooperate
2. Fertile women without sufficient contraceptives
3. Allergy to gabapentin
4. Earlier amputation of the same limb except toes
5. Serious lever, kidney, cardiac, respiratory, haematological disease.-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-05; Study Completion 2006-06

PRIMARY OUTCOMES:
Primary outcome measures:
Number of patients with phantom and stump pain 30 days and 6 months after amputation
Average intensity of stump and phantom pain 30 days and 6 months after amputation

SECONDARY OUTCOMES:
Secondary outcome measures:
Prevalence and severity of phantom and stump pain at controls day 7, 14 and 30, and 3 and 6 months
McGill Pain Questionnaire day 7, 14 and 30, and 3 and 6 months
Concurrent pain medication at day 7, 14 and 30, and 3 and 6 months
Brush evoked allodynia, wind up like pain to repetitive pinprick, pressure pain threshold at day 14 and 30.

CONTACTS AND LOCATIONS:
Overall Officials: Lone Nikolajsen, MD, PhD, Principal Investigator — Danish Pain Research Center
Locations (1):
- Danish Pain Research Center, Aarhus University Hospital, Aarhus, Denmark